CLINICAL TRIAL: NCT01099917
Title: Does Maitake Mushroom Extract Enhance Hematopoiesis in Myelodysplastic Patients? A Phase II Trial
Brief Title: Does Maitake Mushroom Extract Enhance Hematopoiesis in Myelodysplastic Patients?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: YUKIGUNI COMPANY (Unknown); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-094
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; Maitake; mushroom; 09-094
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- Maitake (Experimental): This is a phase II trial examining hematopoietic response in MDS patients.
  Interventions: Drug: Maitake

INTERVENTIONS:
Drug: Maitake — Patients will receive the oral mushroom extract 3mg/kg by mouth twice daily for 3 months. Patients will serve as their own controls, with blood counts after Maitake compared with baseline counts. Rather than a wait list control, at study entry we will obtain from MDS patient charts 2 CBC/differential/platelet values drawn within 12-24 weeks prior to starting the protocol.
  Healthy control volunteers will be recruited to this study as participants for expanding the baseline normal values for neutrophil and monocyte function as measured by the respiratory burst test.

SUMMARY:
Researchers from Memorial Sloan-Kettering Cancer Center, in collaboration with The New York Presbyterian Hospital-Weill Medical College of Cornell University, are conducting a study of a medicinal mushroom extract called Maitake (pronounced my-tock-e).

Laboratory studies show that Maitake can reduce the growth of cancer in animals. The Maitake does not kill cancer cells directly. It is believed to work through the immune system (the body's defense system against infection). Our test tube, animal and human dose determining studies show that Maitake can enhance immune function. We are conducting this study to see whether Maitake improves the neutrophil count and function in patients with MDS. The neutrophils are white blood cells which help to fight infection.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC patients age 18 or older able to sign informed consent
* Absolute Neutrophil count >0.5 K/mcL
* Diagnosis of MDS by bone marrow biopsy
* Patient not a candidate for aggressive standard treatment

Exclusion Criteria:

* IPSS (High risk)
* History of AML
* History of Stem Cell transplant
* Known history of HIV+
* Allergy to mushrooms
* Bone Marrow blasts >10%

HEALTHY CONTROL ELIGIBILTY CRITERIA

Inclusion Criteria

* Age ≥55 years

Exclusion Criteria

* Currently taking corticosteroids or other immunosuppressants
* Known history of HIV+
* Current or previous malignancy or hematology disorder except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Wesa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Maitake: This is a phase II trial examining hematopoietic response in Myelodisplastic Patients.
Period: Overall Study
Arm/Group | Maitake
Started | 45
Completed | 18
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Not Treated | 24

BASELINE CHARACTERISTICS:
Arm/Group | Maitake
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Changes in Neutrophil Counts
Description: The main criterion for study response is ability of the study agent to show a statistically significant improvement in neutrophil count and neutrophil function (as measured by the respiratory burst test). Changes in neutrophil counts will also be described as defined by the International Working Group (IWG) criteria for response in MDS patients
Time Frame: baseline and week 12
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Maitake
Number analyzed (Participants) | 18
cells/mm^3 | -0.3 [-0.5 to 0]

ADVERSE EVENTS:
Arm/Group | Maitake
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maitake (N=21)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aphonia (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maitake (N=21)
Blood bilirubin increased (Blood and lymphatic system disorders) | 2
Headache (General disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 10
Pain in extremity (General disorders) | 2
Platelet count decreased (Blood and lymphatic system disorders) | 9 (9)
White blood cell decreased (Blood and lymphatic system disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes